CLINICAL TRIAL: NCT05569694
Title: Pelvic Health Education for Women in Underserved Communities
Brief Title: Movement-Based Pelvic Health Education for Women in Underserved Communities
Acronym: PHEd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Alexis Kendrick, Assistant Professor of Physical Therapy, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Kendrick PH
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Floor Muscle Weakness; Pelvic Pain
Keywords: Women's health; Community education; Underserved population
MeSH Terms: conditions — Pelvic Pain; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women in the Community (Experimental): Movement-Based pelvic health education
  Interventions: Other: Movement-based pelvic health education

INTERVENTIONS:
Other: Movement-based pelvic health education — A single virtual education session led by a physical therapist trained in pelvic health. The virtual course was approximately one hour and included movement-based education through various positions, exercises, and movements with explanations for each pose as it relates to pelvic health.

SUMMARY:
It is essential to provide the community with evidenced-based care to optimize healthcare outcomes; more specifically, women in underserved communities undergoing health disparities in rehabilitation. To address this issue, a movement-based pelvic health education course was developed to assess women's knowledge and adherence of the exercises in an underserved region in Western Arkansas.The purpose of this research was to determine the effectiveness of a single movement-based pelvic health education session on general pelvic health knowledge, underactive pelvic floor, and overactive pelvic floor knowledge and adherence to performing pelvic exercises in women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* female-identifying
* ability to speak English or provide own translator
* ability to complete the questionnaires
* clearance from physician if pregnant
* access to internet

Exclusion Criteria:

-Experiencing pelvic pain and/or pregnant and does not have physician clearance to participate

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge Acquisition | 1 month
  Participants complete a questionnaire pre, post, and one-month following the intervention. The questionnaire includes true/false questions: 10 general knowledge, 10 underactive pelvic floor, 10 overactive pelvic floor. The more correct answers the participant submits, the higher the score. Answer options: True, False, I don't know.

SECONDARY OUTCOMES:
Exercise Adherence | 1 month
  Participants complete a questionnaire pre-session and one-month following the intervention. The questionnaire included questions related to the number of times per week the participant implemented pelvic floor movements and options were:
  Never less than once a week about once a week 2 or 3 times a week at least once a day twice on most days twice each day

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided